CLINICAL TRIAL: NCT05219643
Title: Effect of Neurally-Adjusted Ventilatory Assist (NAVA) on Weaning Outcome in Patients With Mechanical Ventilation: Multicenter, Single-blind, Parallel, Control, Randomized Clinical Trials
Brief Title: Effect of Nava on Weaning Outcome in Patients With Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Collaborators: First Affiliated Hospital of Wannan Medical College (Other)
Responsible Party: Principal Investigator, Ling Liu, professor, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NAVA2021
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: ARDS
Keywords: NAVA; Weaning; Tracheotomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NAVA (Experimental): Received NAVA.
  Interventions: Device: NAVA
- PSV (Active Comparator): Received PSV.
  Interventions: Device: PSV

INTERVENTIONS:
Device: NAVA — Nava level is set to maintain the target tidal volume: 6-10ml / kg (pbw). The trigger sensitivity is 0.5uv. The expiratory trigger sensitivity: the built-in software of the ventilator is set to 70% of the peak value of diaphragm electrical activity.
  Arms: NAVA
Device: PSV — According to the doctor's experience, maintain the target tidal volume: 6-10ml / kg (pbw); trigger sensitivity: 1.5-2l/min, expiratory trigger sensitivity: 30% inspiratory peak flow rate.
  Arms: PSV

SUMMARY:
This study intends to compare the effects of NAVA and PSV on weaning success rate and mechanical ventilation time in patients with tracheotomy patients through a randomized controlled study.

DETAILED DESCRIPTION:
For patients with difficult weaning, NAVA can shorten the time of mechanical ventilation, but there is no large-scale study to explore the effect of NAVA on the weaning success rate and mechanical ventilation time of patients with gas resection. Therefore, this study intends to compare the effects of NAVA and PSV on weaning success rate and mechanical ventilation time in patients with tracheotomy patients through a randomized controlled study.

It is a prospective, multicenter, parallel group, single blind, randomized controlled tria。

ELIGIBILITY:
Inclusion Criteria:

1. Tracheotomy and invasive mechanical ventilation is expected to be required for > 48h;
2. When support pressure ≤ 15 cmH2O, it can withstand pressure support ventilation (PSV) time > 1h;

Exclusion Criteria:

1. Age < 18 years or > 85 years;
2. Deep sedation.
3. Severe hemodynamic instability (norepinephrine or equivalent converted dose of other vasoactive drugs > 1ug / kg.min or map ≤ 65mmhg)
4. Severe respiratory center depression, high paraplegia, neuromuscular disease;
5. Esophageal obstruction, esophageal perforation, severe esophageal variceal bleeding, upper gastrointestinal surgery, diaphragmatic hernia and thoracic deformity;
6. Patients with chronic respiratory diseases requiring long-term home oxygen therapy;
7. Patients with severe coagulation dysfunction (INR > 1.5, APTT > 44s, history of leukemia);
8. Severe other organ dysfunction is expected to die in a short time (7 days) or palliative treatment.
9. The estimated survival time of advanced solid organ or hematological system tumors is < 30 days
10. Participate in other clinical studies within 30 days;
11. Failing to sign the informed consent form;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
The 28-day ventilator-free days | From enrollment to days 28
  Days alive and free from mechanical ventilation from study drug administration to day 28.

SECONDARY OUTCOMES:
Weaning Success Rate | From enrollment to days 28
  Respective groups weaning Success Rate
Duration of Mechanical Ventilation | From enrollment to days 28.
  Duration of mechanical ventilation within 28 days after enrollment
28-ICU mortality | From enrollment to days 28.
  ICU mortality within 28 days after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Liu Ling, MD, Principal Investigator — Department of Critical Care Medicine, Zhongda Hospital, School of Medicine, Southeast University
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No